CLINICAL TRIAL: NCT03182582
Title: Efficacy of the Er:YAG Laser Debridement on Patient-Reported Pain and Bacterial Load in Chronic Wounds
Brief Title: Efficacy of Laser Debridement on Pain and Bacterial Load in Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Geoffrey C. Gurtner, Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-35141
Record Dates: First submitted 2017-05-31; First posted 2017-06-09 (Actual); Results first posted 2018-04-17 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Wound Open; Chronic Venous Hypertension (Idiopathic) With Ulcer; Diabetic Foot Ulcer
Keywords: Laser Debridement; Debridement
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: A portion of the patients will be randomized to sharp debridement first, then laser for the second debridement. The other portion will undergo this in the opposite order.
Who Masked: Investigator
Masking Description: The investigator is blinded to which patient is receiving sharp or laser debridement as his/her first treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Week 1 - Erbium:Yttrium-Aluminum-Garnet Laser Debridement (Active Comparator): During the first treatment, laser debridement will be performed at 200-um until punctate bleeding is visualized. During the second treatment, sharp debridement will be performed via a scalpel/curette until punctate bleeding is visualized.
  Tissue biopsies will then be obtained from the wounds prior to the first treatment, immediately after the first treatment, immediately prior to the subsequent treatment, and immediately after the second treatment. These will then be sent to Pathogenius for molecular analysis of wound microflora using polymerase chain reaction and sequencing.
  Pain will be assessed during debridement by recording the Numerical Rating Scale for pain assessment.
  Interventions: Device: Erbium:Yttrium-Aluminum-Garnet (Er:YAG) Laser Debridement; Procedure: Scalpel/Curette Debridement
- Week 1 - Scalpel/Curette Debridement (Active Comparator): During the first treatment, sharp debridement will be performed via a scalpel/curette until punctate bleeding is visualized. During the second treatment, laser debridement will be performed at 200-um until punctate bleeding is visualized.
  Tissue biopsies will then be obtained from the wounds prior to the first treatment, immediately after the first treatment, immediately prior to the subsequent treatment, and immediately after the second treatment. These will then be sent to Pathogenius for molecular analysis of wound microflora using polymerase chain reaction and sequencing.
  Pain will be assessed during debridement by recording the Numerical Rating Scale for pain assessment.
  Interventions: Device: Erbium:Yttrium-Aluminum-Garnet (Er:YAG) Laser Debridement; Procedure: Scalpel/Curette Debridement

INTERVENTIONS:
Device: Erbium:Yttrium-Aluminum-Garnet (Er:YAG) Laser Debridement — Laser debridement entailed usage of an Er:YAG laser, employing the JOULE® machine (Sciton, Inc., Palo Alto, California). Full-field ablation was performed using the 2940 nm Er:YAG Contour TRL Resurfacing® application with the following settings: fluence - 50 J/cm2, spot overlap - 50%, pattern repeat - 0.5 seconds, spot size - 3-mm (Figure 1). Debridement was carried out until all fibrinous and/or necrotic tissues were removed, and healthy, bleeding tissue was visualized.
Procedure: Scalpel/Curette Debridement — Using a scalpel/curette, each patient's chronic wound is debrided until healthy, viable tissue is noted.

SUMMARY:
Bacterial load is frequently associated with impaired healing of chronic wounds. As well, sharp debridement is often associated with pain, causing patient distress, and thereby occasionally contributing to inadequacy of debridement, leading to a delay in wound healing. The purpose of this study is to assess the efficacy of the Sciton Laser in reducing bacterial load and patient distress in patients with chronic wounds, in efforts to expedite the wound healing process.

DETAILED DESCRIPTION:
Chronic wounds are a debilitating affliction, affecting a substantial portion of the population worldwide and incurring staggering healthcare economic costs (1,2). Included among chronic wounds are venous leg ulcers, which are known to cause considerable pain, and can impact patient quality of life, thereby complicating wound care (3). The exact pathophysiology and etiology of the prolonged course of chronic wounds are poorly understood, but are thought to be multi-factorial in nature. Given the exposure of chronic wounds to the environment, they harbor a diverse microbial flora. Specifically, there is evidence that biofilm produced by these microbes are a large contributor to their non-healing nature (4). Debridement is considered an integral part of wound management with its ability to remove necrotic tissue and bacterial biofilm, in addition to stimulating release of cytokines and growth factors that promote wound healing (5). However, sharp debridement, the gold standard in wound care, is often ineffective for painful wounds.

The effect of lasers on wound healing have been well-studied both in in vitro and in vivo models. Beneficial effects of low-level laser therapy in wound healing in animal and human studies has been established. However, extrapolation of this data is limited by study design and light dosimetry (6). Laser energy used for surgical excision is a lesser-known debridement technique that has been largely limited to burn scar treatment (7,8,9,10). Lasers are electro-optical devices that emit a focused beam of intense monochromatic light in the visible and infrared radiation spectrums. Since their start in the 1960s, lasers have been successfully utilized in many fields of medicine. Lasers for wound debridement began in the 1970s, with the successful report of a continuous-beam carbon dioxide (CO2) laser used for skin graft preparation of infected decubitus ulcers (11). Laser debridement is based on the controlled vaporization of the superficial layers of the wound bed. This results in the removal of the tissue containing unwanted microbial and necrotic particles. The laser type and the number of passes performed determine the depth of tissue ablation (12). Unlike other methods dependent on the clinician's manual control, laser debridement is electronically controlled, improving precision and reducing the risk of healthy tissue damage. Advantages of laser debridement include precision and uniformity of tissue ablation, which reduces trauma to the wound bed, improving patient comfort. To reduce thermal damage to healthy tissue, several improvements in laser technology have been made over the years. By utilizing a pulsed-beam system, laser energy is delivered in high-power, rapid succession pulses, resulting in short duration and high temperature exposure of target tissue, thereby minimizing thermal injury.

Erbium:YAG (Er:YAG) lasers, with a wavelength of 2940-nm are widely used in the dermatologic community for skin resurfacing, for anti-aging and acne-related purposes (13). Skin ablation with the erbium laser is very precise, and allows for accurate assessment of the resurfacing depth (12,14,15). Since Er:YAG laser energy has greater than twelve times more water absorption efficiency than CO2 lasers, water in the tissue is rapidly expanded to eject the charred debris from the wound surface without leaving behind a necrotic eschar (12,16,17). The Er:YAG laser provides distinct advantages in precise ablation control and the reduction of residual necrotic tissue burden with minimal procedural discomfort, making the Er:YAG laser the most suitable device for laser wound debridement. Preliminary studies demonstrate remarkable patient pain reduction after laser debridement, resulting in more thorough removal of necrotic tissue and biofilm/bacterial load. Additionally, the extent of laser debridement is determined by the laser settings, as opposed to the individual operator's dexterity and skill, thereby providing better control over the wound bed preparation, producing more predictable and reproducible outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged eighteen years or older
* Having a chronic wound (as defined by lack of at least 50% reduction in wound surface area over a period of four weeks)
* No clinical evidence of active wound bed infection
* No exposure of any vital structure (i.e., tendon, bone, vessel)
* Has signed the informed consent form prior to any study protocol related procedure
* Willing and able to adhere to protocol requirements

Exclusion Criteria:

* Any unstable medical condition that would cause the study treatment to be detrimental to the subject, as judged by the Principle Investigator
* Documented medical history of significant cardiac, pulmonary, gastrointestinal, endocrine (other than Diabetes Mellitus type 1 or 2), metabolic, neurological, hepatic or nephrologic disease would impede the subject's participation, as judged by the Principle Investigator
* Documented medical history of immunosuppression, immune deficiency disorder, or currently using immunosuppressive medications
* Having clinical presentation of active osteomyelitis
* Pregnancy or lactation
* Participation in another clinical study involving ulcers within thirty days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Meyer, CCRC, Study Director — Clinical Trial Coordinator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill KE, Davies CE, Wilson MJ, Stephens P, Harding KG, Thomas DW. Molecular analysis of the microflora in chronic venous leg ulceration. J Med Microbiol. 2003 Apr;52(Pt 4):365-369. doi: 10.1099/jmm.0.05030-0. PMID 12676877
- [Background] Collins L, Seraj S. Diagnosis and treatment of venous ulcers. Am Fam Physician. 2010 Apr 15;81(8):989-96. PMID 20387775
- [Background] Palfreyman S. Assessing the impact of venous ulceration on quality of life. Nurs Times. 2008 Oct 14-20;104(41):34-7. PMID 18979958
- [Background] Falanga V. Chronic wounds: pathophysiologic and experimental considerations. J Invest Dermatol. 1993 May;100(5):721-5. doi: 10.1111/1523-1747.ep12472373. No abstract available. PMID 8491995
- [Background] Brem H, Stojadinovic O, Diegelmann RF, Entero H, Lee B, Pastar I, Golinko M, Rosenberg H, Tomic-Canic M. Molecular markers in patients with chronic wounds to guide surgical debridement. Mol Med. 2007 Jan-Feb;13(1-2):30-9. doi: 10.2119/2006-00054.Brem. PMID 17515955
- [Background] Percival SL, Francolini I, Donelli G. Low-level laser therapy as an antimicrobial and antibiofilm technology and its relevance to wound healing. Future Microbiol. 2015;10(2):255-72. doi: 10.2217/fmb.14.109. PMID 25689537
- [Background] Evison D, Brown RF, Rice P. The treatment of sulphur mustard burns with laser debridement. J Plast Reconstr Aesthet Surg. 2006;59(10):1087-93. doi: 10.1016/j.bjps.2006.02.010. Epub 2006 Jul 7. PMID 16996434
- [Background] Graham JS, Schomacker KT, Glatter RD, Briscoe CM, Braue EH Jr, Squibb KS. Efficacy of laser debridement with autologous split-thickness skin grafting in promoting improved healing of deep cutaneous sulfur mustard burns. Burns. 2002 Dec;28(8):719-30. doi: 10.1016/s0305-4179(02)00198-5. PMID 12464469
- [Background] Lam DG, Rice P, Brown RF. The treatment of Lewisite burns with laser debridement---'lasablation'. Burns. 2002 Feb;28(1):19-25. doi: 10.1016/s0305-4179(01)00078-x. PMID 11834325
- [Background] Reynolds N, Cawrse N, Burge T, Kenealy J. Debridement of a mixed partial and full thickness burn with an erbium:YAG laser. Burns. 2003 Mar;29(2):183-8. doi: 10.1016/s0305-4179(02)00247-4. No abstract available. PMID 12615469
- [Background] Stellar S, Meijer R, Walia S, Mamoun S. Carbon dioxide laser debridement of decubitus ulcers: followed by immediate rotation flap or skin graft closure. Ann Surg. 1974 Feb;179(2):230-7. doi: 10.1097/00000658-197402000-00022. No abstract available. PMID 4590105
- [Background] Alster TS, Lupton JR. Erbium:YAG cutaneous laser resurfacing. Dermatol Clin. 2001 Jul;19(3):453-66. doi: 10.1016/s0733-8635(05)70286-2. PMID 11599402
- [Background] Pozner JN, Goldberg DJ. Superficial erbium:YAG laser resurfacing of photodamaged skin. J Cosmet Laser Ther. 2006 Jun;8(2):89-91. doi: 10.1080/14764170600717852. PMID 16766487
- [Background] Bass LS. Erbium:YAG laser skin resurfacing: preliminary clinical evaluation. Ann Plast Surg. 1998 Apr;40(4):328-34. doi: 10.1097/00000637-199804000-00002. PMID 9555984
- [Background] Weinstein C. Computerized scanning erbium:YAG laser for skin resurfacing. Dermatol Surg. 1998 Jan;24(1):83-9. doi: 10.1111/j.1524-4725.1998.tb04058.x. PMID 9464295
- [Background] Weinstein C, Pozner J, Scheflan M, Achauer BM. Combined Erbium:YAG Laser Resurfacing and Face Lifting. Plast Reconstr Surg. 2001 Feb;107(2):593-594. doi: 10.1097/00006534-200102000-00046. No abstract available. PMID 11242368
- [Background] Roberts TL 3rd, Pozner JN. Lasers, facelifting, and the future. Clin Plast Surg. 2000 Apr;27(2):293-9. No abstract available. PMID 10812528
- Available data/document: Study Protocol — https://eprotocol.stanford.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser, Then Sharp: During the first treatment, laser debridement will be performed at 200-um until punctate bleeding is visualized. During the second treatment, sharp debridement will be performed via a scalpel/curette until punctate bleeding is visualized.
  Tissue biopsies will then be obtained from the wounds prior to the first treatment, immediately after the first treatment, immediately prior to the subsequent treatment, and immediately after the second treatment. These will then be sent to Pathogenius for molecular analysis of wound microflora using polymerase chain reaction and sequencing.
  Pain will be assessed during debridement by recording the Numerical Rating Scale for pain assessment.
- Sharp, Then Laser: During the first treatment, sharp debridement will be performed via a scalpel/curette until punctate bleeding is visualized. During the second treatment, laser debridement will be performed at 200-um until punctate bleeding is visualized.
  Tissue biopsies will then be obtained from the wounds prior to the first treatment, immediately after the first treatment, immediately prior to the subsequent treatment, and immediately after the second treatment. These will then be sent to Pathogenius for molecular analysis of wound microflora using polymerase chain reaction and sequencing.
  Pain will be assessed during debridement by recording the Numerical Rating Scale for pain assessment.
Period: Treatment 1
Arm/Group | Laser, Then Sharp | Sharp, Then Laser
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0
Period: Treatment 2
Arm/Group | Laser, Then Sharp | Sharp, Then Laser
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Laser and Sharp Debridement: Laser debridement will be performed at 200-um until punctate bleeding is visualized. Sharp debridement will be performed via a scalpel/curette until punctate bleeding is visualized.
  Tissue biopsies will then be obtained from the wounds prior to the first treatment, immediately after the first treatment, immediately prior to the subsequent treatment, and immediately after the second treatment. These will then be sent to Pathogenius for molecular analysis of wound microflora using polymerase chain reaction and sequencing.
  Pain will be assessed during debridement by recording the Numerical Rating Scale for pain assessment.
Arm/Group | Laser and Sharp Debridement
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22
Wound Etiology [Count of Participants; unit: Participants]
  Diabetic | 4
  Venous | 11
  Other | 7
Wound size [Mean (Standard Deviation); unit: cm] | 3.6 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Pain With Debridement
Description: Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is used in our study to measure the intensity or frequency of pain. We have used Numerical Rating Scale (NRS), variant of VAS, which is a validated, uni-dimensional measure of pain intensity reported on an 11-point numeric scale. The scores were reported from "0" to "10," with "0" representative of "no pain," and "10" representative of the "worst possible pain".
Time Frame: Day 1 of the respective procedure (immediately following)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Laser Debridement: Laser debridement was performed at 200-um until punctate bleeding is visualized. Pain was assessed during debridement by recording the Numerical Rating Scale for pain assessment.
- Sharp Debridement: Sharp debridement was performed via a scalpel/curette until punctate bleeding is visualized. Pain was assessed during debridement by recording the Numerical Rating Scale for pain assessment.
Arm/Group | Laser Debridement | Sharp Debridement
Number analyzed (Participants) | 22 | 22
units on a scale | 3.0 (1.7) | 4.8 (2.6)
Statistical Analysis 1: Comparison: Laser Debridement vs Sharp Debridement; A sample size of 22 patients was required to achieve 80% power, using a two-tailed test with α = 0.05; Test type: Superiority; p = 0.003, Paired t test

2. Primary Outcome: Bacterial Load Pre- and Post-Laser Debridement
Description: Bacterial load in wound as per tissue biopsy, pre- and post-laser debridement. CFU = Colony Forming Units.
Time Frame: Day 1 of the laser procedure (immediately before and after)
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Laser Debridement: A tissue biopsy was performed prior to laser debridement. This tissue was analyzed for bacterial load.
- Post-Laser Debridement: A tissue biopsy was performed after laser debridement. This tissue was analyzed for bacterial load.
Arm/Group | Pre-Laser Debridement | Post-Laser Debridement
Number analyzed (Participants) | 22 | 22
Participants
  Negative | 0 | 2
  <10^5 CFU/g | 6 | 11
  >=10^5 CFU/g | 16 | 9

3. Primary Outcome: Bacterial Load Pre- and Post-Sharp Debridement
Description: Bacterial load in wound as per tissue biopsy, pre- and post-sharp debridement
Time Frame: Day 1 of the sharp procedure (immediately before and after)
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Sharp Debridement: A tissue biopsy was performed prior to curette/scalpel debridement. This tissue was analyzed for bacterial load.
- Post-Sharp Debridement: A tissue biopsy was performed after curette/scalpel debridement. This tissue was analyzed for bacterial load.
Arm/Group | Pre-Sharp Debridement | Post-Sharp Debridement
Number analyzed (Participants) | 22 | 22
Participants
  Negative | 0 | 5
  <10^5 CFU/g | 12 | 10
  >=10^5 CFU/g | 10 | 7

4. Secondary Outcome: Patient Preference
Description: Patient-reported preference of debridement type one week after study completion, reported as the count of participants that preferred either method.
Time Frame: 2 weeks
Population: Survey respondents were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Laser and Sharp Debridement
Number analyzed (Participants) | 17
Participants
  Prefer laser | 9
  Prefer sharp | 6
  Unsure | 2

5. Secondary Outcome: Percent Change in Wound Size- Immediately Post-debridement
Description: The mean wound size increased immediately after debridement in both Groups, compared to the mean wound size before the debridement.
Time Frame: Day 1 of the respective procedure (immediately after)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Laser Debridement | Sharp Debridement
Number analyzed (Participants) | 22 | 22
percent change | 40.2 (95.0) | 63.4 (96.8)

6. Secondary Outcome: Percent Change in Wound Size - 1 Week Post-debridement
Description: The mean percent change in wound size 1-week post-laser debridement was -20.8% ± 80.1%, as compared with -36.7% ± 54.3% 1-week post-sharp debridement (p = 0.6).
Time Frame: 1 week following respective procedure
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Laser Debridement | Sharp Debridement
Number analyzed (Participants) | 22 | 22
percent change | -20.8 (80.1) | -36.7 (54.3)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks
Arm/Group | Laser Debridement | Sharp Debridement
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

LIMITATIONS AND CAVEATS:
4 different surgeons carried out wound debridement and tissue sampling; therefore, techniques could vary in wound bed preparation and tissue sampling. Also, wound measurements suffer from variations in technique and inter-observer subjectivity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03182582/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT03182582/SAP_001.pdf